CLINICAL TRIAL: NCT01068457
Title: Chronic Pain After Thoracotomy (VATS)
Brief Title: Chronic Pain After Thoracotomy (Video Assisted Thoracic Surgery - VATS)
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: MD Kim Wildgaard, Section for Surgical Pathophysiology 4074
Other Study IDs: VATS-hb2008-059
Record Dates: First submitted 2010-02-08; First posted 2010-02-15 (Estimated); Last update posted 2010-07-14 (Estimated); Status verified 2010-07

CONDITIONS: Neuropathic Pain; Thoracic Surgery, Video Assisted; Chronic Pain
Keywords: persistent pain; neuropathic pain; Thoracic Surgery, Video Assisted; Chronic Pain
MeSH Terms: conditions — Neuralgia; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PTPS: Patients with pain after VATS
- Pain free: Patients reporting no pain late after VAT

SUMMARY:
This is an explorative study investigating potential nerve injury after VATS.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and give consent
* Can read
* Residing in Denmark

Exclusion Criteria:

* Unable to understand the written information in Danish
* Abuse (Medicine, Drugs, Alcohol)
* Severe psychiatric Illness
* Conflicting neurological disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Thresholds via QST | Late postoperatively (3months)

CONTACTS AND LOCATIONS:
Locations (1):
- Section for Surgical Pathophysiology 4074 andSection of Acute Pain management and Palliative Medicine., Copenhagen, Denmark

REFERENCES:
- [Background] Wildgaard K, Ravn J, Kehlet H. Chronic post-thoracotomy pain: a critical review of pathogenic mechanisms and strategies for prevention. Eur J Cardiothorac Surg. 2009 Jul;36(1):170-80. doi: 10.1016/j.ejcts.2009.02.005. PMID 19307137